CLINICAL TRIAL: NCT04691596
Title: Promoting Contextually Cued Physical Activity Habits: A Pilot Study Using Cue-Contingent Financial Incentives for Daily Walking
Brief Title: Promoting Contextually Cued PA Habits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Chad Stecher@asu.edu, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1698
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Exercise
Keywords: Physical activity; Financial incentives; mHealth
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were randomized into four different study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Active Comparator): One fourth of participants were assigned to the Control Group, and received a basic training with the StepUp app and were asked to contact the study team with any problems or questions they encountered during the eight-week study period. No other intervention tools or app reminders were provided to the Control Group.
  Interventions: Behavioral: App use instructions
- Treatment Group 1 (Experimental): Additionally eligible to receive weekly $5 Amazon gift cards over the first four weeks of the study for performing a ≥10-minute walk (i.e. non-cue-contingent incentives)
  Interventions: Behavioral: Non-cue-contingent weekly incentives; Behavioral: App use instructions
- Treatment Group 2 (Experimental): Received an instructional video on the benefits of contextual-cue-dependent habits and instructions on how to identify an optimal personalized cue that would consistently trigger their ≥10-minute walking habit, then they were similarly eligible weekly for $5 Amazon gift cards over the first four weeks conditional on completing a ≥10-minute walk at any time of day (i.e. non-cue-contingent incentives)
  Interventions: Behavioral: Non-cue-contingent weekly incentives; Behavioral: Habit Coaching; Behavioral: App use instructions
- Treatment Group 3 (Experimental): Received an instructional video on the benefits of contextual-cue-dependent habits and instructions on how to identify an optimal personalized cue that would consistently trigger their ≥10-minute walking habit, then they were eligible weekly for $5 Amazon gift cards over the first four weeks conditional on completing a ≥10-minute walk at any the pre-specified time of their chosen contextual cue (i.e. cue-contingent incentives)
  Interventions: Behavioral: Cue-contingent weekly incentives; Behavioral: Habit Coaching; Behavioral: App use instructions

INTERVENTIONS:
Behavioral: Non-cue-contingent weekly incentives — Eligible to win $5 Amazon gift card conditional on completing a daily ≥10-minute walk at any time of day
  Arms: Treatment Group 1; Treatment Group 2
Behavioral: Cue-contingent weekly incentives — Eligible to win $5 Amazon gift card conditional on completing a daily ≥10-minute walk within a +/-1 hour window of the pre-specified time of their chosen contextual walking cue
  Arms: Treatment Group 3
Behavioral: Habit Coaching — Received an instructional video on the benefits of contextual-cue-dependent habits and instructions on how to identify an optimal personalized cue that would consistently trigger their ≥10-minute walking habit
  Arms: Treatment Group 2; Treatment Group 3
Behavioral: App use instructions — Received a basic training with the StepUp app

SUMMARY:
The primary goal of this two-month pilot study is to measure the behavioral change induced by targeted habit formation reminders that are surfaced via an iPhone app and financial incentives that were offered conditional on using a personalized contextual cue for a daily walking habit. The data and user feedback collected during this study will also be used to optimize the design and content of the iPhone app, which will be tested in future, larger scale experimental research.

DETAILED DESCRIPTION:
Subjects for this research are recruited on campus at Rensselaer Polytechnic Institute and the State University of New York at Albany, and their participation was incentivized. After meeting the eligibility criterion (including have at least some intrinsic motivation for increasing physical activity), downloading the project's iPhone app, and signing the project consent form, all participants will have their step count data recorded for an 8-week study period.

Existing interventions that have successfully improved study participants' health-related behaviors typically find that behavioral changes do not persist beyond 3 months after the intervention period. Fortunately, novel habit formation interventions from the psychology literature offer the potential for building long-term behavioral change and avoiding the common "relapse triangles" observed in these existing behavioral interventions. These new methods are based on the theory that habits are formed through the repetition of the same behavior in response to a stable, environmental cue. After an initial period of repetition, automaticity is formed, and the behavioral response becomes more effortlessly/unconsciously induced by the environmental cue. Behavioral reminders that reinforce a specific behavioral routine-environmental cue pair have been shown to support this initial period of habit formation; however, given the individualized nature of these reminders, a generalizable intervention method has not been developed and empirically tested. This research will use an iPhone app to examine the role of both general informational on contextually cued habits and the use of personalized reminders and financial incentives for using a daily physical activity contextual cue on the persistence of physical activity behavior after the intervention tools are withdrawn.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* Have an existing wellness goal related to increasing physical activity
* Access to an iPhone with iOS 10 or above (in order to use the app)
* Proficiency in speaking and reading English

Exclusion Criteria:

* Have a major visual impairment
* Pregnancy
* Expected surgery
* A chronic or acute health condition that affects their ability to perform basic mobility tasks or light-aerobic exercise (e.g. heart disease, injured or missing limb, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2020-08-21 (Actual)

PRIMARY OUTCOMES:
Daily Step Count | 8 weeks
  Full study period analyses
Daily Step Count | 4 weeks
  Follow-up period

SECONDARY OUTCOMES:
Habitual daily walking | 8 weeks
  Whether walking occurred within +/- 1 hour of contextual cue; full study period
Habitual daily walking | 4 weeks
  Whether walking occurred within +/- 1 hour of contextual cue; follow-up period
10,000 daily step | 4 weeks
  Likelihood of reaching 10,000 daily steps, follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Rensselaer Polytechnic Institute, Troy, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stawarz, Cox, and Blandford. 2015. "Beyond self-tracking and reminders: designing smartphone apps that support habit formation." Proceedings of the 33rd annual ACM conference on human factors in computing systems, ACM.
- [Background] Lally, Phillippa, et al. 2010. "How are habits formed: Modelling habit formation in the real world." European journal of social psychology 40(6): 998-1009.
- [Background] Wood W, Neal DT. A new look at habits and the habit-goal interface. Psychol Rev. 2007 Oct;114(4):843-63. doi: 10.1037/0033-295X.114.4.843. PMID 17907866
- [Background] Wood and Neal. 2016. "Healthy through habit: Interventions for initiating & maintaining health behavior change." Behavioral Science & Policy 2(1): 71-83.
- [Background] Adriaanse MA, Gollwitzer PM, De Ridder DT, de Wit JB, Kroese FM. Breaking habits with implementation intentions: a test of underlying processes. Pers Soc Psychol Bull. 2011 Apr;37(4):502-13. doi: 10.1177/0146167211399102. Epub 2011 Feb 11. PMID 21317315
- [Derived] Stecher C, Chen CH, Codella J, Cloonan S, Hendler J. Combining anchoring with financial incentives to increase physical activity: a randomized controlled trial among college students. J Behav Med. 2024 Oct;47(5):751-769. doi: 10.1007/s10865-024-00492-4. Epub 2024 May 5. PMID 38704776